CLINICAL TRIAL: NCT06987955
Title: Evaluation of Clinical Success of Bioactive and Fluoride Resin Based Pit and Fissure Sealants: A Split Mouth Clinical Study
Brief Title: Clinical Evaluation of Pit and Fissure Sealants
Status: Completed | Type: Observational
Sponsor: Canan Bayraktar Nahir (Other)
Collaborators: Tokat Gaziosmanpasa University (Other)
Responsible Party: Sponsor-Investigator, Canan Bayraktar Nahir, Assistant Professor, Tokat Gaziosmanpasa University
Organization: Tokat Gaziosmanpasa University (Other)
Other Study IDs: 23-KAEK-150
Record Dates: First submitted 2025-05-07; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Pit and Fissure Sealants
Keywords: children; BioCoat; Fissurit FX; modified USPHS
MeSH Terms: conditions — Van der Woude syndrome | interventions — Pit and Fissure Sealants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mandibular right first molar
  Interventions: Other: Biocoat Pit and fissure sealant
- Mandibular right left molar
  Interventions: Other: Fissurit FX Pit and fissure sealant

INTERVENTIONS:
Other: Biocoat Pit and fissure sealant — Application of Biocoat
  Groups: Mandibular right first molar
Other: Fissurit FX Pit and fissure sealant — Application of Fissurit FX
  Groups: Mandibular right left molar

SUMMARY:
Pit and fissure sealants are considered an effective preventive approach in protecting teeth from caries, particularly by transforming deep, plaque-retentive occlusal surfaces into smooth, easily cleanable areas. These materials act as a physical barrier on the tooth surface, limiting the access of microorganisms to nutrients and thereby inhibiting bacterial activity. In this thesis study, the long-term clinical performance of a newly introduced bioactive resin-based pit and fissure sealant, BioCoat™ (Premier, USA), was compared with that of a fluoride-releasing resin-based sealant, Fissurit FX (Voco, Germany). The null hypothesis of the study was that there would be no statistically significant difference in the clinical success rates between the two sealant materials.

DETAILED DESCRIPTION:
This study was designed to evaluate the clinical effectiveness of BioCoat™ (Premier, USA), a newly introduced bioactive resin-based pit and fissure sealant, and Fissurit FX (Voco, Germany), a fluoride-releasing resin-based sealant, in children aged 7 to 9 years who presented to the Department of Pedodontics at the Faculty of Dentistry, Tokat Gaziosmanpaşa University.

Sealants were applied to the mandibular first permanent molars (teeth 36 and 46) of 63 patients using a split-mouth design. Group 1 received the bioactive material BioCoat™ (Premier, USA), while Group 2 was treated with the fluoride-releasing resin Fissurit FX (Voco, Germany). The sealants were evaluated over an 18-month period based on the modified United States Public Health Service (USPHS) criteria.

The modified USPHS criteria assess parameters including marginal discoloration, marginal adaptation, retention, and the presence of secondary caries in fissure sealant materials. Each parameter is scored as alpha, bravo, or charlie. While alpha and bravo scores indicate clinical success, the presence of a charlie score in any parameter is considered indicative of treatment failure. In clinical follow-ups, cases with one or more charlie (C) scores were classified as unsuccessful, the sealant was replaced, and these cases were excluded from further analysis.

Statistical analysis was performed using IBM SPSS Statistics version 23 (IBM Corp., Armonk, NY, USA). Cochran's Q test was employed to compare intra-group clinical success rates across different time points.

ELIGIBILITY:
Inclusion Criteria:

Parental consent obtained Cooperative behavior rating of 3 or 4 according to the Frankl Behavior Rating Scale Requirement for non-invasive pit and fissure sealant application Age between 7 and 9 years

Exclusion Criteria:

Presence of mental or physical disability History of allergy to any medication or dental restorative material Presence of parafunctional habits Cooperative behavior rating of 1 or 2 according to the Frankl Behavior Rating Scale

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 7-9 years old who apply to Tokat Gaziosmanpaşa University, Faculty of Dentistry, Department of Pedodontics.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of 18-month clinical success of pit and fissure sealants | 18 month
  Comparison of the clinical performance of pit and fissure sealants over an 18-month period based on modified USPHS criteria (marginal adaptation, marginal discoloration, retention, and the presence of secondary caries).
  Note: The modified USPHS criteria assess parameters including marginal discoloration, marginal adaptation, retention, and the presence of secondary caries in pit anf fissure sealant materials. Each parameter is scored as alpha, bravo, or charlie. While alpha and bravo scores indicate clinical success, the presence of a charlie score in any parameter is considered indicative of treatment failure. In clinical follow-ups, cases with one or more charlie (C) scores were classified as unsuccessful, the sealant was replaced, and these cases were excluded from further analysis.

SECONDARY OUTCOMES:
Comparison of the intraoral survival rates of pit and fissure sealants | 18 month
  Comparative evaluation of the cumulative survival curves of pit and fissure sealants over an 18-month follow-up period using Kaplan-Meier analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanapaş University, Tokat Province, Kaleardı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
with the link to be prepared later

REFERENCES:
- [Background] Abdelsalam, A. F., Haridy, M. F., Hamza, H. S. E., Farid, M. R., & Shaalan, O. O. (2022). Clinical evaluation of bioactive resin based pits & fissures sealants versus conventional resin based pits & fissures sealants in caries susceptible fissures in permanent molars: A randomized controlled. International Journal of Health Sciences, 6(S7), 2745-2759. Abdelsalam, A. F., Haridy, M. F., Hamza, H. S. E., Farid, M. R., & Shaalan, O. O. (2022). Clinical evaluation of bioactive resin based pits & fissures sealants versus conventional resin based pits & fissures sealants in caries susceptible fissures in permanent molars: A randomized controlled. International Journal of Health Sciences, 6(S7), 2745-2759.
- See also: Clinical evaluation of bioactive resin based pits & fissures sealants versus conventional resin based pits & fissures sealants in caries susceptible fissures in permanent molars: A randomized controlled. — https://sciencescholar.us/journal/index.php/ijhs/article/view/12039